CLINICAL TRIAL: NCT03047356
Title: Effects of "If-then" Plans ("Implementation Intentions") on Adolescent Sleep
Brief Title: Sleep Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Christopher Armitage, Professor of Health Psychology, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Carding_1
Record Dates: First submitted 2017-02-03; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Mental

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First-person "if-then" plan (Experimental): Participants are asked to form "if-then" plans and the instructions are presented in the first person ("if I...then I..."). "Ifs" are critical situations, "thens" are appropriate responses.
  Interventions: Behavioral: "If-then" plans
- Second-person "if-then" plan (Experimental): Participants are asked to form "if-then" plans and the instructions are presented in the second person ("if you...then you..."). "Ifs" are critical situations, "thens" are appropriate responses.
  Interventions: Behavioral: "If-then" plans
- Control (Placebo Comparator): Participants are presented with "ifs "(critical situations) and "thens" but are not asked to form "if-then" plans.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: "If-then" plans — "If-then" plans (or "implementation intentions") involve linking in memory critical situations (e.g., temptations) with appropriate responses (e.g., substitution)
  Arms: First-person "if-then" plan; Second-person "if-then" plan
Other: Control — Exposure to critical situations (e.g., temptations) and appropriate responses (e.g., substitution) but not linked in memory
  Arms: Control

SUMMARY:
A trial that tests whether implementation intentions improve sleep among adoelescents.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-16 years

Exclusion Criteria:

* Unable or unwilling to complete the question

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-06 (Actual)

PRIMARY OUTCOMES:
Achieving recommended sleep levels | 1 month
  The main outcome measure was adapted from the Pittsburgh Sleep Quality Index (Buysse, Reynolds, Monk, Berman, & Kupfer, 1989), and was designed to tap both quantity and quality of sleep. Sleep quantity was assessed by asking: "How many hours of actual sleep do you normally get on a night before school? _________ hours," "What time do you normally go to bed on a night before school? __________ pm," and "What time do you normally get up on a school day? __________ am."

SECONDARY OUTCOMES:
Self-regulation | 1 month
  Sniehotta, Nagy, and Scholz's (2006) six items were used to capture three facets of action control (Karoly, 1993) on 7-point (+1 to +7) strongly disagree-strongly agree scales. (e.g., "During the last month I constantly monitored my sleep on the nights before school")
Habit | 1 month
  Gardner et al.'s (2012) self-report behavioral automaticity index, which consists of four items measured on 7-point strongly disagree-strongly agree scales. The items are: "Getting 9 hours' sleep on the nights before school is something I do automatically," "Getting 9 hours' sleep on the nights before school is something I do without thinking," "Getting 9 hours' sleep on the nights before school is something I do without having to consciously remember," and "Getting 9 hours' sleep on the nights before school is something I start doing before I realize I'm doing it."

IPD SHARING:
Plan to Share IPD: Undecided